CLINICAL TRIAL: NCT04273035
Title: The Effect of Handheld-multimedia Versus Oral Midazolam Preanesthetic on the Level of Perioperative Anxiety in Pediatric Day-care Surgery: A Randomized Controlled Trial
Brief Title: Handheld-multimedia Versus Oral Midazolam in Pediatric on Perioperative Anxiety
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/318; 2019-004671-39 (EudraCT Number)
Record Dates: First submitted 2020-02-05; First posted 2020-02-17 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Perioperative Anxiety; Preanesthetic Medication; Inhalation Anesthesia; Ambulatory Surgery; Tonsillectomy; Circumcision; Dental Care
Keywords: Preanesthetic medication; Handheld computer; Midazolam; Multimedia; Anxiety; Mask induction; Day Care Surgery
MeSH Terms: conditions — Anxiety Disorders | interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: Group A: midazolam premedicated, standard of care Group B: IPAD, no midazolam premedication
Masking Description: digital block randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Midazolam Group (Active Comparator): * Midazolam(Buccolam 5mg/ml)
  * 0.5mg/kg oral, max 12mg
  * one time
  * given 30 min prior to going to holding
  Interventions: Drug: Midazolam oral solution
- IPAD group (Active Comparator): * No premedication
  * IPAD when arriving at the holding
  * any games, movies, clips, puzzles
  Interventions: Device: IPAD

INTERVENTIONS:
Drug: Midazolam oral solution — Oral Buccolam
  Other Names: Buccolam
  Arms: Midazolam Group
Device: IPAD — Playing any game, film, clip or puzzle on a tablet till after induction of anesthesia
  Other Names: Handheld multimedia, tablet
  Arms: IPAD group

SUMMARY:
The first goal of this study is to compare the efficacy and safety between anxiolysis by multimedia-distraction with an IPAD versus anxiolysis by premedication with midazolam prior to the induction. Secondly to evaluate the need for midazolam-premedication in pediatric day-care patients induced by inhalational anesthesia.

DETAILED DESCRIPTION:
Perioperative anxiety in children is a common multifactorial influenced and triggered entity with an incidence as high as 50%. Especially (mask)induction of anesthesia is considered one of the most stressful experiences for a child undergoing surgery. A common practice worldwide to diminish the level of anxiety prior to anesthesia is premedication with the benzodiazepine midazolam in order to improve cooperation during induction.

Premedication with midazolam has a primary purpose to reduce preoperative anxiety and has inherent to a benzodiazepine its sedative effects. Although these effects are implied, negative effects of premedication: respiratory complications, paradoxical negative behavior has been reported. Although alternative medications have been studied, studies for non-pharmacological anxiety-reduction remain limited.

Non-pharmacological anxiety-reduction by distraction including Tablet or IPAD-multimedia might be a readily available alternative for midazolam premedication. Potentially limiting the use of psychoactive agents, limiting the need for preoperative sedation and therefore possibly decrease secondary respiratory complications in pediatric surgical day-care.

Objective:

The first goal of this study is to compare the efficacy and safety between anxiolysis by multimedia-distraction with an IPAD versus anxiolysis by premedication with midazolam prior to the mask-induction of anesthesia. Secondly to evaluate the need for midazolam premedication in pediatric day-care surgery patients induced by inhalational anesthesia.

ELIGIBILITY:
Inclusion criteria

* Age ≥ 1 year and <8 years old
* ASA class 1 or 2 (American Society of Anesthesiologists Physical Status Classification System)
* Elective circumcision, tonsillectomy or adenoidectomy, dental care procedure in day-care
* Written informed consent by the legal parents or caretaker

Exclusion criteria

* Parents of the patient wish not to participate with the study
* Parents are not able to give informed consent (language barrier, legally incapable)
* A contraindication for the use of premedication with midazolam
* A known allergy to midazolam
* A contraindication for premedication in general
* A contraindication for the use of a gas-induction/gas-anesthesia
* A contraindication for the use of sevoflurane
* A known mental retardation of the child
* Preoperative behavioral disturbances and psychiatric disorders
* Any use of psychoactive medication
* A known photosensitive epilepsy
* A previous operation within 3 months of the time of scheduled operation
* Any other contraindication for the use of the study medication
* Previous history of multiple surgery (>3)

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Anxiety level at induction | Directly prior to induction of anesthesia, 20 minutes
  Measured bij Short version modified Yale Preoperative Anxiety Scale(mYPAS-SF), scoring activity 1-4/4, vocalizations 1-6/6, emotional expressivity 1-4/4, state of apparent arousal 1-4/4, parental use 1-4/4, subtotal is the sum of all the individual scores divided by their number of choices, mYpas-SF total score is subtotal/5 * 100 and therefore a score between 23,3-100 Scored prior moment of mask induction (T2)
Anesthesiologist Satisfaction Induction | During induction of anesthesia 10 minutes
  Satisfactory Score for Induction/Anesthesia: 5 point scale: Very satisfactory, Satisfactory, Neutral, Unsatisfactory and Very satisfactory Scored in the OR directly post induction

SECONDARY OUTCOMES:
Anxiety level at Daycare | Leaving daycare, 10 minutes
  Measured bij Short version modified Yale Preoperative Anxiety Scale(mYPAS-SF), scoring activity 1-4/4, vocalizations 1-6/6, emotional expressivity 1-4/4, state of apparent arousal 1-4/4, parental use 1-4/4, subtotal is the sum of all the individual scores divided by their number of choices, mYpas-SF total score is subtotal/5 * 100 and therefore a score between 23,3-100 Scored at Daycare (T0) when leaving to holding
Anxiety level at holding | On holding, 20 minutes
  Measured bij Short version modified Yale Preoperative Anxiety Scale(mYPAS-SF), scoring activity 1-4/4, vocalizations 1-6/6, emotional expressivity 1-4/4, state of apparent arousal 1-4/4, parental use 1-4/4, subtotal is the sum of all the individual scores divided by their number of choices, mYpas-SF total score is subtotal/5 * 100 and therefore a score between 23,3-100 Scored at holding (T1) 10 minutes after arrival
Anxiety level at recovery | 15 minutes after awake, 30 minutes
  Measured bij Short version modified Yale Preoperative Anxiety Scale(mYPAS-SF), scoring activity 1-4/4, vocalizations 1-6/6, emotional expressivity 1-4/4, state of apparent arousal 1-4/4, parental use 1-4/4, subtotal is the sum of all the individual scores divided by their number of choices, mYpas-SF total score is subtotal/5 * 100 and therefore a score between 23,3-100 Scored at recovery (T3) 15 minutes after awake
Anxiety level Change Daycare vs OR | change during daycare (T0) and induction(T2) in the OR, average 1 hour
  Measured bij Short version modified Yale Preoperative Anxiety Scale(mYPAS-SF), scoring activity 1-4/4, vocalizations 1-6/6, emotional expressivity 1-4/4, state of apparent arousal 1-4/4, parental use 1-4/4, subtotal is the sum of all the individual scores divided by their number of choices, mYpas-SF total score is subtotal/4 * 100 and therefore a score between 23,3-100
Sedation level at Daycare | 10 minutes
  Richmond Agitation-Sedation Scale, RASS-score between -5 till + 4 Scored at Daycare (T0) when leaving to holding
Sedation level at holding | 20 minutes
  Richmond Agitation-Sedation Scale, RASS-score between -5 till + 4 Scored (T1) 10 minutes after arrival holding
Sedation level at induction | 10 minutes
  Richmond Agitation-Sedation Scale, RASS-score between -5 till + 4 Scored at moment of mask induction (T2)
Sedation level at recovery | 30 minutes
  Richmond Agitation-Sedation Scale, RASS-score between -5 till + 4 Scored 15 minutes after arrival recovery (T3)
Laryngospasm at induction | 10 minutes
  Laryngospasm by Four-point scale:
  1. No Laryngospasm
  2. Mild laryngospasm (relieved by jaw thrust and 100% oxygen),
  3. Moderate laryngospasm (relieved by 100% oxygen and positive pressure ventilation)
  4. Severe laryngospasm (relieved by succinylcholine and intubation) Scored in the OR post-induction
Laryngospasm post extubation/post laryngeal mask | 10 minutes
  Laryngospasm by Four-point scale:
  1. No Laryngospasm
  2. Mild laryngospasm (relieved by jaw thrust and 100% oxygen),
  3. Moderate laryngospasm (relieved by 100% oxygen and positive pressure ventilation)
  4. Severe laryngospasm (relieved by succinylcholine and intubation) Scored in the OR post detubation/post laryngeal mask
Bronchospasm postinduction | 10 minutes
  Bronchospasm/wheezing 1. Yes 2. No • In absence of scale Scored in the OR postinduction
Bronchospasm post detubation/laryngeal mask | 10 minutes
  Bronchospasm/wheezing 1. Yes 2. No • In absence of scale Scored in the OR post detonation/laryngeal mask
Postoperative Pain | 40 minutes
  The pain observation scale for young children (POCIS-Score) score 0-7, scoring 0 or1 for • face-expression: frowning/grimaces = 1, sound crying/moan =1, breathing: irregular/gasping/holding=1, body tonus: tense/shiver/restless =1, movement of arms: tense/fist/restless =1, movement of legs: tense/pulled up/flexed = 1, mood: agitation/restless = 1 Scored on the recovery 30 minutes after arrival
Parental Satisfaction on the anxiety-management at daycare | 10 minutes
  1. Very satisfied
  2. Satisfied
  3. Neutral
  4. Unsatisfactory
  5. Very Unsatisfactory Scored at daycare-surgery (T0)
Parental Satisfaction on the anxiety-management at holding | 10 minutes
  1. Very satisfied
  2. Satisfied
  3. Neutral
  4. Unsatisfactory
  5. Very Unsatisfactory Scored at holding (T1)
Parental Satisfaction on the anxiety-management at OR | 10 minutes
  1. Very satisfied
  2. Satisfied
  3. Neutral
  4. Unsatisfactory
  5. Very Unsatisfactory Scored after induction and parent has left the OR (T2)
Parental Satisfaction on the anxiety-management at recovery | 10 minutes
  1. Very satisfied
  2. Satisfied
  3. Neutral
  4. Unsatisfactory
  5. Very Unsatisfactory Scored at the recovery (T3)
Parental Stress level at day care | 10 minutes
  Parental Stress level in 5 - point scale- ´I feel':
  1. Extremely Stressed
  2. Very stressed
  3. moderate stressed
  4. Low stressed
  5. Very low stressed scored at day care (T0)
Parental Stress level at holding | 10 minutes
  Parental Stress level in 5 - point scale- ´I feel':
  1. Extremely Stressed
  2. Very stressed
  3. moderate stressed
  4. Low stressed
  5. Very low stressed Scored at holding (T1)
Parental Stress level at OR | 10 minutes
  Parental Stress level in 5 - point scale- ´I feel':
  1. Extremely Stressed
  2. Very stressed
  3. moderate stressed
  4. Low stressed
  5. Very low stressed Scored at OR (T2)
Parental Stress level at recovery | 10 minutes
  Parental Stress level in 5 - point scale- ´I feel':
  1. Extremely Stressed
  2. Very stressed
  3. moderate stressed
  4. Low stressed
  5. Very low stressed Scored at recovery (T3)
Overall Parental Satisfaction | 10 minutes
  5- Point scale
  1. Very satisfied
  2. Satisfied
  3. Neutral
  4. Unsatisfactory
  5. Very Unsatisfactory Scored when leaving recovery
Child Stress level by parent at daycare | 10 minutes
  Child Stress level by parent, 5- Point scale
  1. Happy, plays
  2. Slightly worried
  3. Worried, stops playing
  4. Fears, crying
  5. Hysterical Scored at daycare-surgery (T0)
Child Stress level by parent at holding | 10 minutes
  Child Stress level by parent, 5- Point scale
  1. Happy, plays
  2. Slightly worried
  3. Worried, stops playing
  4. Fears, crying
  5. Hysterical Scored at holding (T1)
Child Stress level by parent at OR | 10 minutes
  Child Stress level by parent, 5- Point scale
  1. happy, plays
  2. slightly worried
  3. worried, stops playing
  4. fear, crying
  5. hysterical Scored at OR after induction (T2)
Child Stress level by parent at Recovery | 10 minutes
  Child Stress level by parent, 5- Point scale
  1. Happy, plays
  2. Slightly worried
  3. Worried, stops playing
  4. Fear, crying
  5. Hysterical Scored at recovery (T3)

OTHER OUTCOMES:
Postoperative need for pain medication | 1 hour
  Postoperative need for pain medication, indicated as yes or no, and description of medication with given dose Noted on the recovery
Postoperative need for anti-nausea/vomiting medication | 1 hour
  Postoperative need for anti-nausea/vomiting medication, indicated as yes or no, and description of product with given dose Noted on the recovery
Time arrival recovery to time leaving recovery | 2 hour
  Time arrival recovery to time leaving recovery, time notation on arrival and leaving Noted on the recovery

CONTACTS AND LOCATIONS:
Overall Officials: Alex Van Hoorn, MD, Principal Investigator — Resident of department of Anesthesiology
Locations (1):
- Universitair Ziekenhuis Brussel (UZ Brussel), Jette, Belgium

IPD SHARING:
Plan to Share IPD: Yes
* Individual participant data will be available after deidentification
  * For researchers who provide a methodological proposal
  * Achieving aims in the proposal
  * Proposals needs to be directed to the principal investigators
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available 3 months after study publication for 10 years
Access Criteria: Written request and providing a methodological proposal